CLINICAL TRIAL: NCT04231565
Title: Study on Therapeutic Effects and Safety of Nucleoside (Acid) Analogues Treatment in Patients With Chronic Hepatitis B With Normal Alanine Aminotransferase and Positive Hepatitis B Virus DNA: a Randomized Controlled Trial
Brief Title: Nucleoside (Acid) Analogues Treatment in Patients With Normal ALT and Positive HBVDNA.
Acronym: ALTHBV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL10
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis B Virus
Keywords: hepatitis B virus; nucleoside; nucleotide
MeSH Terms: conditions — Hepatitis B | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAF group (Active Comparator): 100 patients would receive treatment of oral Tenofovir alafenamide Fumarate(TAF) 25 mg once per day from baseline to life-long unless the patient achieves HBsAg loss.
  Interventions: Drug: Tenofovir alafenamide Fumarate
- Observation group (No Intervention): 100 patients would not receive treatment from baseline to life-long.

INTERVENTIONS:
Drug: Tenofovir alafenamide Fumarate — Patients would receive treatment of oral Tenofovir alafenamide Fumarate（TAF）once per day.
  Other Names: Vemlidy
  Arms: TAF group

SUMMARY:
This study is to investigate the clinical efficacy and safety of Nucleoside (acid) analogues treatment in patients with normal Alanine Aminotransferase and positive Hepatitis B virus DNA.

DETAILED DESCRIPTION:
Hepatitis b virus infection has always been a global public health problem that endangers national health. Current clinical guidelines do not recommend antiviral therapy for people with positive hepatitis b-DNA and normal Alanine Aminotransferase, but studies have found that viral replication is associated with an increased risk of cirrhosis and liver tumors. Nucleoside (acid) analogues can effectively inhibit viral reverse transcriptase, reduce HBV viral load in the blood, thereby reducing secondary inflammation, and contribute to liver cell regeneration and disease recovery. And its side effect is small, adverse reaction rate is low, use safety.

ELIGIBILITY:
Inclusion Criteria:

* Positive hepatitis b surface antigen and hepatitis b antibody > 0.5 year;
* Age from 18 to 65 years old;
* Serum Alanine Aminotransferase(ALT) ≤1×ULN at least 12 weeks;
* Positive Hepatitis b virus(HBV);
* Do not receive nucleotide/nucleoside analogues or interferon treatment in the past half year.

Exclusion Criteria:

* Other active liver diseases;
* Hepatocellular carcinoma or other malignancy;
* Pregnancy or lactation;
* Human immunodeficiency virus infection or congenital immune deficiency diseases; 5.Severe diabetes, autoimmune diseases; 6.Other important organ dysfunctions; 7.Using glucocorticoid; 8.Patients can not follow-up; 9.Investigator considering inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
hepatitis b s antigen decrease from baseline | 48 week, 96 week, 144 week
  Magnitude of decrease in hepatitis B antigen quantification from baseline to week 144.

SECONDARY OUTCOMES:
hepatitis b e antigen loss rate | 48 week, 96 week, 144 week
  Hepatitis b e antigen would be tested to know the ratio of patients with negative hepatitis B e antigen.
hepatitis b virus(HBV) DNA undetectable rate | 48 week, 96 week, 144 week
  Hepatitis b virus DNA would not be detected if it below the upper limit of test value
hepatitis b virus(HBV) RNA undetectable rate | 48 week, 96 week, 144 week
  Hepatitis b virus RNA would not be detected if it below the upper limit of test value
hepatitis b s antigen loss rate | 48 week, 96 week, 144 week
  Hepatitis b s antigen become negative and quantitative analysis below the upper limit of test value

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article (text, tables, figures and appendices) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following the article publication.
Access Criteria: Proposals should be directed to xxx@yyy. To gain access, data requestors need to sign a data access agreement.

REFERENCES:
- [Derived] Luo Q, Xu W, Zhang Y, Li X, Lai J, Li J, Zheng X, Deng H, Chen L, Zhu X, Xie C, Peng L. Tenofovir Alafenamide Fumarate Reduces Virological Replication in HBeAg-Negative Patients With Normal Alanine Aminotransferase: A 48-Week Randomised Controlled Trial. J Viral Hepat. 2026 Mar;33(3):e70141. doi: 10.1111/jvh.70141. PMID 41608776
- [Derived] Wang L, Zhu S, Liu Y, Zheng L, Xu W, Luo Q, Zhang Y, Deng H, Li X, Xie C, Peng L. Prognostic value of decline in model for end-stage liver disease score and hepatic encephalopathy in hepatitis B-related acute-on-chronic liver failure patients treated with plasma exchange. Scand J Gastroenterol. 2022 Sep;57(9):1089-1096. doi: 10.1080/00365521.2022.2063032. Epub 2022 Apr 17. PMID 35435091
- [Derived] Wang L, Xu W, Li X, Chen D, Zhang Y, Chen Y, Wang J, Luo Q, Xie C, Peng L. Long-term prognosis of patients with hepatitis B virus-related acute-on-chronic liver failure: a retrospective study. BMC Gastroenterol. 2022 Apr 2;22(1):162. doi: 10.1186/s12876-022-02239-4. PMID 35366805
- [Derived] Wang L, Wu L, Li X, Zhang Y, Lai J, Zhu X, Xie C, Peng L. Tenofovir alafenamide fumarate therapy in subjects with positive HBV-DNA and normal levels of alanine transaminase: a study protocol for a randomised controlled trial. BMJ Open. 2021 Aug 18;11(8):e048410. doi: 10.1136/bmjopen-2020-048410. PMID 34408049